CLINICAL TRIAL: NCT06923449
Title: Gastric Cancer' Textbook Oncological Outcome and Tumor Board Performance - The Experience of a High-volume Italian University Hospital
Brief Title: Gastric Cancer' Textbook Oncological Outcome and Tumor Board Performance
Acronym: GaC-TOP
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Società Italiana di Chirurgia Oncologica SICO - ESSO affiliated (Unknown)
Responsible Party: Sponsor
Other Study IDs: ID 6671 Prot.n.0010178/24
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Stomach Neoplasm
Keywords: Gastric Cancer; Multidisciplinary Tumor Board; Textbook Outcome; Textbook Oncological Outcome
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-TB: All subsequent patients aged 18 years or older, surgical candidates with curative intent, with a pathology-confirmed diagnosis of gastric adenocarcinoma, treated at Fondazione Policlinico Universitario Agostino Gemelli IRCCS of Rome from jan 2018 to november 2019
- Post-TB: All subsequent patients aged 18 years or older, surgical candidates with curative intent, with a pathology-confirmed diagnosis of gastric adenocarcinoma, treated at Fondazione Policlinico Universitario Agostino Gemelli IRCCS of Rome from december 2019 onwards
  Interventions: Other: Multidisciplinary Tumor Board

INTERVENTIONS:
Other: Multidisciplinary Tumor Board — Institution of Multidisciplinary Tumor Board for Gastric Cancer at Fondazione Policlinico Gemelli in november 2019
  Groups: Post-TB

SUMMARY:
The goal of this observational, no-profit, spontaneous, retrospective, monocentric study is to compare surgical and oncologic outcomes in patients affected by gastric cancer before and after the institution of the Tumor Board, a multidisciplinary weekly case discussion. The main question it aims to answer is whether the Textbook Outcome (TO) and Textbook Oncological Outcome (TOO) of patients with non-early, non-metastatic gastric cancer undergoing surgical treatment with curative intent have improved before (from January 2018 to November 2019) and after (from December 2019 onwards) the establishment of the Multidisciplinary Tumor Board (MTB) at Fondazione Policlinico Gemelli (FPG).

DETAILED DESCRIPTION:
Background. Textbook Outcome (TO) is a composite parameter for quality in surgical oncology proposed by the Dutch Upper Gastrointestinal Cancer Audit (DUCA) group, directly related to survival [1]. A Polish group proposed an integration to the TO, adding the item perioperative chemotherapy administration compliance (POC), for a comprehensive assessment of multimodal treatment in gastric cancer (GaC) patients' management, named Textbook Oncological Outcome (TOO) [2]. This has been subsequently validated in the European GASTRODATA database [3], showing a correlation with lower 90-day mortality rates. The latter study acknowledges a TO of 68.5%, higher than previous experiences reported from the Western world, while reporting a TOO of only 22.8%, pointing out the need to improve multimodal treatment of GC patients.

To evaluate any influence of systematic Multidisciplinary Tumor Board (MTB) on patient outcomes, we aim to assess TO, TOO, Time from first diagnosis To first Therapy (TTT), the appropriateness of Patient to Treatment Allocation (PTA), and MTB hospital Adherence (TBA) as indicators of Tumor Board Performance (TBP) before and after its institution. At Policlinico Universitario Agostino Gemelli, the MTB for GaC was established in November 2019. We will collect data from 2018 to date in order to minimize bias due to different perioperative regimens.

Hypothesis. We hypothesize a global improvement in GaC patients' TO and TOO following the institution of the MTB.

Objectives. The study's primary objective is to evaluate the Textbook Outcome (TO) and Textbook Oncological Outcome (TOO) of patients with gastric cancer undergoing surgical treatment with curative intent before (from January 2018 to November 2019) and after (from December 2019 onwards) the establishment of the Multidisciplinary Tumor Board (MTB) at Fondazione Policlinico Gemelli (FPG) (primary endpoint: percentage of patients achieving TO and TOO out of the total number of patients who underwent surgery with curative intent for gastric cancer at FPG before and after the MTB institution). Secondary objectives include assessing Tumor Board Performance (TBP) by measuring: - Time from diagnosis To Treatment, the interval between diagnosis and beginning of the first oncological treatment (TTT; endpoint: delay in days/weeks from diagnosis to treatment before and after MTB institution), - Patient to Treatment Allocation (PTA; endpoint: percentage of upfront surgery candidates who do not receive adjuvant chemotherapy before and after MTB institution) and - Tumor Board Adherence (TBA; endpoint: percentage of patients operated on at FPG who were previously discussed at the MTB out of the total number of patients who underwent surgery with curative intent for gastric cancer at FPG).

Methods. We will review clinical, pathological, surgical and oncological data of patients affected by Gastric Cancer candidated for surgical intervention -either upfront, either post neoadjuvant treatment, either in conversion surgery- with curative intent for primary and secondary outcomes.

Expected results. This study aims to demonstrate an improvement in Gastric Cancer patients' outcomes, such as Textbook Outcome (TO) and Textbook Oncological Outcome (TOO), following the establishment of the MTB. Additionally, we anticipate enhanced Tumor Board Performance over time, thanks to the improvements of Time from Diagnosis to Treatment (TTT), Tumor Board Adherence (TBA), and Patient to Treatment Allocation (PTA), attributable to a learning effect.

ELIGIBILITY:
Inclusion Criteria:

* pathology-confirmed diagnosis of gastric adenocarcinoma
* age 18 years or older
* surgical candidates with curative intent

Exclusion Criteria:

* Endoscopic Mucosal Resection (EMR) or Endoscopic Submucosal Dissection (ESD)
* previous EMR or ESD (salvage surgery)
* histologies other than adenocarcinoma (no squamous cell carcinomas, GISTs, sarcomas, lymphomas, etc)
* unsufficient staging (unclear clinical stage at diagnosis)
* emergency presentation (obstrucetd, significantly bleeding, perforated gastric cancer)
* synchronous tumors affecting survival
* pregnant patients
* age <18years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subsequent patients aged 18 years or older, surgical candidates with curative intent, with a pathology-confirmed diagnosis of gastric adenocarcinoma, treated at Fondazione Policlinico Universitario Agostino Gemelli IRCCS of Rome from 2018 to date.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Textbook Outcome (TO) | january 2018 - february 2024
  fulfillment of 10 items consisting in (1) radical resection according to the surgeons' assessment at the end of the operation, (2) no intraoperative complications, (3) negative resection margins (R0), (4) at least 15 lymph nodes (LNs) retrieved and examined, (5) no severe postoperative complications, (6) no reinterventions, (7) no readmission to intensive care unit (ICU), (8) no prolonged hospital stay (21 days), (9) no postoperative mortality, and (10) no hospital readmission
Textbook Oncologic Outcome (TOO) | january 2018 - february 2024
  TOO is defined by the addition of PeriOperative Chemotherapy (POC) or Adjuvant chemoTherapy (AT) administration to the 10 TO items resulting in 11 items

SECONDARY OUTCOMES:
Time To first Treatment (TTT) | january 2018 - february 2024
  TTT is defined as the interval from diagnosis to first treatment (first chemotherapy administration or radical surgery), the diagnosis will be traced to the date of final pathology of endoscopic biopsies; TTT will be subdivided in Staging Time (ST), time from first histology to completion of staging, and Waiting list Time (WT), time from last staging exam to first treatment
Patient to Treatment Allocation (PTA) | january 2018 - february 2024
  PTA appropriateness, indicated by the percentage of newly diagnosed patients undergoing upfront surgery who are not offered adjuvant therapy. This may be due to either early staging or because the patient is deemed unfit for systemic treatment. PTA will be calculated in patients aged 80y or younger, given that older patients less frequently receive neoadjuvant chemotherapy
Tumor Board Adherence (TBA) | january 2018 - february 2024
  TBA expressed as the percentage of patients who undergo surgery for Gastric Cancer at FPG after being discussed at the MTB over the totality of patients surgically treated for GaC at FPG

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Biondi, Prof., Principal Investigator — Fondazione Policlinico Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, IT, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busweiler LA, Schouwenburg MG, van Berge Henegouwen MI, Kolfschoten NE, de Jong PC, Rozema T, Wijnhoven BP, van Hillegersberg R, Wouters MW, van Sandick JW; Dutch Upper Gastrointestinal Cancer Audit (DUCA) group. Textbook outcome as a composite measure in oesophagogastric cancer surgery. Br J Surg. 2017 May;104(6):742-750. doi: 10.1002/bjs.10486. Epub 2017 Feb 27. PMID 28240357
- [Background] Sedlak K, Rawicz-Pruszynski K, Mlak R, Geca K, Skorzewska M, Pelc Z, Malecka-Massalska T, Polkowski WP. Union is strength: Textbook outcome with perioperative chemotherapy compliance decreases the risk of death in advanced gastric cancer patients. Eur J Surg Oncol. 2022 Feb;48(2):356-361. doi: 10.1016/j.ejso.2021.08.005. Epub 2021 Aug 11. PMID 34404560
- [Background] Sedlak K, Rawicz-Pruszynski K, Mlak R, Van Sandick J, Gisbertz S, Pera M, Dal Cero M, Baiocchi GL, Celotti A, Morgagni P, Vittimberga G, Hoelscher A, Moenig S, Kolodziejczyk P, Richter P, Gockel I, Piessen G, Da Costa PM, Davies A, Baker C, Allum W, Romario UF, De Pascale S, Rosati R, Reim D, Santos LL, D'ugo D, Wijnhoven B, Degiuli M, De Manzoni G, Kielan W, Frejlich E, Schneider P, Polkowski WP. Textbook Oncological Outcome in European GASTRODATA. Ann Surg. 2023 Nov 1;278(5):823-831. doi: 10.1097/SLA.0000000000006054. Epub 2023 Aug 9. PMID 37555342
- [Background] Pillay B, Wootten AC, Crowe H, Corcoran N, Tran B, Bowden P, Crowe J, Costello AJ. The impact of multidisciplinary team meetings on patient assessment, management and outcomes in oncology settings: A systematic review of the literature. Cancer Treat Rev. 2016 Jan;42:56-72. doi: 10.1016/j.ctrv.2015.11.007. Epub 2015 Nov 24. PMID 26643552
- [Background] Hanna TP, King WD, Thibodeau S, Jalink M, Paulin GA, Harvey-Jones E, O'Sullivan DE, Booth CM, Sullivan R, Aggarwal A. Mortality due to cancer treatment delay: systematic review and meta-analysis. BMJ. 2020 Nov 4;371:m4087. doi: 10.1136/bmj.m4087. PMID 33148535
- [Background] Kim TH, Suh YS, Huh YJ, Son YG, Park JH, Yang JY, Kong SH, Ahn HS, Lee HJ, Slankamenac K, Clavien PA, Yang HK. The comprehensive complication index (CCI) is a more sensitive complication index than the conventional Clavien-Dindo classification in radical gastric cancer surgery. Gastric Cancer. 2018 Jan;21(1):171-181. doi: 10.1007/s10120-017-0728-3. Epub 2017 Jun 8. PMID 28597328
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Pak LM, Yang T, Wang J. The safety and efficacy of gastrectomy for gastric cancer among octogenarians: a western population-based study. J Geriatr Oncol. 2019 Jul;10(4):598-603. doi: 10.1016/j.jgo.2018.10.012. Epub 2018 Oct 24. PMID 30366851